CLINICAL TRIAL: NCT06521073
Title: The Effect of Traınıng on Paın, Actıvıtıes of Daıly Lıfe and Patıent Satısfactıon in Patıents Who Had Total Knee Prosthesıs
Brief Title: Educatıon in Patıents Who Had Total Knee Prosthesıs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, İlknur tura, Research Assistant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06.01.2024/129
Record Dates: First submitted 2024-06-14; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Prosthesis-Related Infections; Pain, Postoperative; Analgesia
Keywords: education; pain; Total Knee Prosthesis
MeSH Terms: conditions — Prosthesis-Related Infections; Pain, Postoperative; Agnosia; Pain | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Before Surgery HBF ONE SAO Patient Education Material Post-Operation (1st, 2nd, 3rd day) ONE SAO Patient Education Material 10-14. BI and PSA will be applied on days and 6 weeks.
  Interventions: Behavioral: education
- Control (No Intervention): Before Surgery HBF ONE SAO Routine verbal training of the clinic Post-Operation (1st, 2nd, 3rd day) ONE SAO Routine verbal training of the clinic 10-14. BI and PSA will be applied on days and 6 weeks.

INTERVENTIONS:
Behavioral: education — Patient Information Form (HBF): This form, prepared by scanning the literature, includes the patient's age, gender, marital status, education level, profession, social security, place of residence, presence of caregivers in the family, from whom he/she receives care, chronic diseases, the side on which knee prosthesis is applied, knee prosthesis. It is a form consisting of questions about your training status, who you received your training from, and your satisfaction with the training.
  Barthel Index (BI): Barthel activities of daily living index is an evaluation scale used to measure an individual's performance in daily living activities. The index is used for activities of daily living in 10 domains. The Turkish validity and reliability of the Barthel index, developed by Barthel and Mahoney (1965), was determined by Küçükdeveci et al. (17).
  Arms: Experimental

SUMMARY:
The main purposes of nursing care and education for patients who will undergo total knee prosthesis are; The aim is to reduce pain, prevent complications that may develop due to orthopedic surgery, increase patient satisfaction, and preserve function and mobilization.

DETAILED DESCRIPTION:
The knee joint is one of the largest joints in the body and is responsible for maintaining mobilization. This joint is treated with surgery in cases where medical treatment and physiotherapy are ineffective and pain and loss of function increase. For this reason, degenerative diseases of the knee joint are mostly treated with Total Knee Prosthesis (TKA) surgery. TKA is a surgical intervention that reconstructs the joint in patients with knee osteoarthritis, in order to reduce pain and regain lost functions in cases where there is no response to conservative treatment.

TKA is applied to patients whose daily activities are restricted due to pain, limitation of movement, deformity and instability and who cannot achieve the expected improvement with conservative treatment methods (2-4). However, after TKA, life-threatening physical and functional problems and complications that reduce the quality of life and such as pain, infection, pretibial edema, deterioration in bowel functions, pulmonary embolism (PE), deep vein thrombosis (DVT) and prosthesis dislocation may develop.

Early diagnosis and treatment of physical and psychological problems that may occur in these patients, and provision of qualified training that supports patients; self-care competence and functions will accelerate the recovery process and increase the quality of life and patient satisfaction. In a study evaluating health care needs in the early period after TKA. Regarding reducing the pain of patients before discharge, rehabilitation exercises, wound monitoring and care; It has been determined that there is an expectation to be informed about the problems that may occur after discharge, things to pay attention to in the home environment, activities that should not be done, and check-up times.

The main purposes of nursing care and education for patients who will undergo total knee prosthesis are; The aim is to reduce pain, prevent complications that may develop due to orthopedic surgery, increase patient satisfaction, and preserve function and mobilization. It is the nurses duty to determine the patients needs, help the patient when necessary, and ensure continuity of care in cooperation with the patient, his family and the healthcare team. For this reason, nursing care should support the patient and his family until they are equipped with the necessary strength, desire and knowledge, and in this way, individuals should help the patient and their family to gain their independence as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* 18 age over
* Being literate,
* Having knee replacement surgery for the first time;
* Not having chronic diseases or psychiatric diagnoses that would delay wound healing,
* Except hypertension;
* İt will include not developing any early complicationsthe research was planned to be carried out in three stages.

Exclusion Criteria:

* Hospitalized for at least 24 hours
* Agreeing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 1 week
  Patient Information Form (PIF) This form, prepared by scanning the literature, includes the patient's age, gender, marital status, education level, profession, social security, place of residence, presence of caregivers in the family, from whom he/she receives care, chronic diseases, the side on which knee prosthesis is applied, knee prosthesis. It is a form consisting of questions about your training status, who you received your training from, and your satisfaction with the training.

SECONDARY OUTCOMES:
Secondary Outcome Measures | 12 weeks
  Barthel Index (BI):
  Barthel activities of daily living index is an evaluation scale used to measure an individual's performance in daily living activities. The index is used for activities of daily living in 10 domains. This scale, which questions nutrition, washing, self-care, dressing, bowel control, bladder control, toilet use, the ability to move from a wheelchair to a bed and vice versa, mobility and going up and down stairs, consists of a total of 10 items rated on a 0-15 point scale. In this scale, where the possible score ranges from 0 to 100, the high score means the degree to which the individual can function independently (0-20 points are fully dependent, 21-61 points are highly dependent, 62-90 points are moderately dependent, 91-99 points are mildly dependent). dependent, 100 points completely independent).

OTHER OUTCOMES:
Third Outcome Measures | 12 weeks
  Numerical Pain Scale (NRS):
  It is used in patients with scale awareness. 0: I have no pain; 10: indicates unbearable pain and is frequently used in pain assessment in conscious patients. Patients indicate the degree of pain they experience on a scale of 0 to 10; 0 represents no pain and 10 represents the worst possible pain. Thanks to this scale, the patient indicates the worst and mildest pain level he has experienced in the last 24 hours (source).

CONTACTS AND LOCATIONS:
Overall Officials: sevban arslan, Study Director — Cukurova Universty

IPD SHARING:
Plan to Share IPD: No